CLINICAL TRIAL: NCT00043849
Title: Treatment of Agitation/Psychosis in Dementia/Parkinsonism (TAP/DAP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IA0034
Record Dates: First submitted 2002-08-14; First posted 2002-08-15 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2006-08

CONDITIONS: Dementia; Parkinson Disease
Keywords: Psychosis; Agitation, Psychomotor
MeSH Terms: conditions — Dementia; Parkinson Disease; Psychotic Disorders; Psychomotor Agitation | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine

SUMMARY:
The primary aim of this study is to determine the safety and efficacy of quetiapine (Seroquel) for the treatment of psychosis and/or agitation in patients with primary dementia complicated by coexistent parkinsonism, or patients with Parkinson's disease with dementia [PDD] who have episodes of agitation or psychosis. The secondary aim is to determine the safety and tolerability, particularly the influence on parkinsonism, of quetiapine when used to treat psychosis and/or agitation in patients with dementia complicated by coexistent parkinsonism.

DETAILED DESCRIPTION:
Psychosis and agitation often occur in the course of dementia and are a major source of patient disability and caregiver stress. For the common situation in which extrapyramidal (parkinsonian) motor dysfunction accompanies dementia, there is a therapeutic dilemma since the most frequently used drugs to treat the behavioral problems, neuroleptic antipsychotics, can worsen parkinsonism and have been associated with severe extrapyramidal reactions in some types of dementia. To date, the efficacy and tolerability of a promising alternative medication class to treat psychosis and agitation, namely atypical antipsychotics, has not been tested in patients with a primary dementia selected for coexisting parkinsonism.

This is a multicenter double-blind, controlled clinical trial in which 60 subjects with a primary dementia (probable Alzheimer's disease [AD] or probable dementia with Lewy bodies [DLB]) and coexisting parkinsonism, or Parkinson's disease with dementia [PDD] will be randomized to 1 of 2 treatment groups: (1) quetiapine (QUET); an atypical antipsychotic with a favorable extrapyramidal side effect profile), or (2) placebo. Each subject participates in the trial for 10 weeks and systematic ratings of behavior, motor function, cognition, adverse events and other outcomes occur at baseline and after 6 and 10 weeks of assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English or Spanish.
* Presence of dementia as defined by the Diagnostic and Statistical Manual of Psychiatry, 4th ed. (DSM-IV) American Psychiatric Association. 1994.
* Meets NINDS/ADRDA diagnostic criteria for probable Alzheimer's disease [AD] or Consortium diagnostic criteria for probable dementia with Lewy bodies [DLB] or diagnostic criteria for Parkinson's disease with dementia [PDD].
* Presence of psychosis and/or agitation that interferes with daily activities: a) psychosis, b) hallucination, c) delusion, or d) agitation.
* Presence of 2 or more of the following extrapyramidal motor features: a) resting tremor, b) bradykinesia, c) limb rigidity, d) shuffling, short-stepped gait.
* Sum of ratings for the resting tremor, bradykinesia, rigidity and gait items of the Unified Parkinson's Disease Rating Scale (UPDRS) motor examination component must be greater than or equal to 2.
* Brief Psychiatric Rating Scale (BPRS) score greater than or equal to 12.
* Informed consent by participant or an appropriate proxy.
* Spouse/caregiver who is willing and able to accompany the subject to all clinic visits.
* A stable dosage of non-excluded medications for at least 2 weeks prior to the Screening Visit.
* Is in a stable medical condition for at least 4 weeks prior to the Screening Visit.
* Physically acceptable for this study as confirmed by medical history, physical exam and clinical laboratory tests.
* Must be able to ingest oral medications.
* Supervision must be available for administration of study medication.
* Taking any marketed cholinesterase inhibitor (donepezil [Aricept], rivastigmine [Exelon], galantamine [Reminyl], tacrine [Cognex], and/or memantine at a dose unchanged for at least 2 weeks prior to the screening visit.
* Participants may reside in their own home or in a supervised care setting, such as a nursing home.

Exclusion Criteria:

* Mini Mental Status Examination Score <8.
* Use of any of the following in the 3 weeks prior to the screening visit: (a) a neuroleptic or atypical antipsychotic medication; or (b) an anticholinergic drug, amantadine for the treatment of parkinsonism [treatment with levodopa (Sinemet, Sinemet CR) and any dopamine agonist, selegiline or entacapone is allowed].
* A history of a severe adverse reaction to any antipsychotic medication.
* A serious medical illness that would preclude the safe administration of quetiapine, including active cancer. Skin tumors other than malignant melanoma are not exclusionary. Patients with stable prostate cancer may be included at the discretion of the Program Director.
* Current evidence or history in the last 2 years of epilepsy, focal brain lesion, head injury with loss of consciousness and/or immediate confusion after the injury.
* Known pregnancy.

Excluded Medications During the Study:

* Any classical neuroleptic antipsychotic, such as haloperidol (Haldol).
* Any atypical antipsychotic, such as risperidone (Risperidal), quetiapine (Seroquel), ziprasidone (Geodon), olanzapine (Zyprexa) and clozapine (Clozaril).
* Any anxiolytic other than lorazepam (Ativan), as described above. This includes clonazepam (Klonopin), diazepam (Valium), oxazepam (Serax), clorazepate (Tranxene), buspirone (Buspar) and hydroxyzine (Vistaril).
* Any hypnotic other than lorazepam (Ativan), as described above. This includes estazolam (Prosom), flurazepam (Dalmane), quazepam (Doral), temazepam (Restoril), triazolam (Halcion), diphenhydramine (Benadryl), doxylamine (Unisom), zolpidem (Ambien), zaleplon (Sonata) and chloral hydrate.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-07; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Kurlan, MD, Principal Investigator — University of Rochester Medical Center, Department of Neurology
Locations (21):
- United States (21):
  - University of Alabama at Birmingham, Alzheimer's Disease Research Center, Birmingham, Alabama
  - University of California, San Diego, Alzheimer's Disease Center, La Jolla, California
  - VA Healthcare System Long Beach, Long Beach, California
  - University of California at Los Angeles, Alzheimer's Disease Center, Los Angeles, California
  - Stanford/VA Aging Clinical Research Center, Department of Psychiatry & Behavioral Sciences, Palo Alto, California
  - Emory University, Alzheimer's Disease Center, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Southern Illinois University, School of Medicine, Springfield, Illinois
  - E. N. Rogers Memorial Veterans Hospital, Bedford, Massachusetts
  - University of Nevada, Las Vegas, Nevada
  - Parkinson's Disease and Movement Disorders Center, Albany Medical College, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Columbia University, Alzheimer's Disease Research Center, New York, New York
  - University of Rochester Medical Center, Alzheimer's Disease Center, Rochester, New York
  - Syracuse VA Medical Center, Syracuse, New York
  - University of Pittsburgh, Alzheimer's Disease Research Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center at Dallas, Alzheimer's Disease Center, Dallas, Texas
  - Memory Clinic at Southwestern Vermont Medical Center, Bennington, Vermont
  - Fletcher Allan Health Care, Inc., Burlington, Vermont
  - University of Washington at Seattle, Alzheimer's Disease Research Center, Seattle, Washington

REFERENCES:
- [Background] Cummings JL, Knopman D. Advances in the treatment of behavioral disturbances in Alzheimer's disease. Neurology. 1999 Sep 22;53(5):899-901. doi: 10.1212/wnl.53.5.899. No abstract available. PMID 10496242
- [Background] Ballard C, Grace J, McKeith I, Holmes C. Neuroleptic sensitivity in dementia with Lewy bodies and Alzheimer's disease. Lancet. 1998 Apr 4;351(9108):1032-3. doi: 10.1016/s0140-6736(05)78999-6. No abstract available. PMID 9546516
- [Background] McManus DQ, Arvanitis LA, Kowalcyk BB. Quetiapine, a novel antipsychotic: experience in elderly patients with psychotic disorders. Seroquel Trial 48 Study Group. J Clin Psychiatry. 1999 May;60(5):292-8. PMID 10362435